CLINICAL TRIAL: NCT00816647
Title: A Prospective Randomized Study of Medial Patellofemoral Ligament Reconstruction Compared With Medial Reefing
Brief Title: A Prospective Randomized Study of Medial Patellofemoral Ligament (MPFL) Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped for benefit of the MPFL reconstruction arm and due to safety concerns of the medial reefing arm.
Sponsor: Finnish Defense Forces (Other Government)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Petri Sillanpaa, M.D., Tampere University Hospital, Department of Musculosceletal Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPFL08
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2009-07

CONDITIONS: Patella-Dislocation; Patellofemoral Osteoarthritis; Patellar Instability
Keywords: Patella; Dislocation; Knee; Medial Patellofemoral Ligament
MeSH Terms: conditions — Patellar Dislocation; Patella Fracture; Joint Dislocations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Medial patellofemoral ligament reconstruction
  Interventions: Procedure: Patellofemoral stabilizing surgery
- 2 (Active Comparator): Medial reefing
  Interventions: Procedure: Patellofemoral stabilizing surgery

INTERVENTIONS:
Procedure: Patellofemoral stabilizing surgery — Comparison of surgical techniques

SUMMARY:
The operative management of chronic patellar instability has been controversial. Medial patellofemoral ligament reconstruction has gained success recently and might be superior to other soft-tissue procedures. The objective of this prospective study was to compare the clinical outcome after medial patellofemoral ligament reconstruction compared with medial reefing for chronic patellar instability.

DETAILED DESCRIPTION:
Many of the previous studies on medial patellofemoral ligament (MPFL) reconstruction for patellar instability have been difficult to interpret, either because the study setting has included both first-time and recurrent dislocations, or because a lack of control group. Moreover, several studies have enrolled patients with a wide age range, and the majority of the studies have employed retrospective and nonrandomized study designs. Therefore the investigators designed a prospective, randomized study with the primary goal to compare the outcome after MPFL reconstruction with medial reefing for chronic patellar instability. The distance between tibial tubercle and trochlear groove is measured on MRI and corrected if it exceeds 17mm. Primary outcome measure is the occurrence of recurrent objective and subjective patellar instability. The second goal is to evaluate the development of articular cartilage lesions within the patellofemoral joint, and assess clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Chronic patellar instability (more than 2 dislocations)
* Minimum 6 months nonoperative treatment

Exclusion Criteria:

* Severe PF OA
* Acute patellar dislocation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Recurrent patellar instability | 2 years

SECONDARY OUTCOMES:
Patellofemoral osteoarthrosis progression. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Petri J Sillanpaa, M.D., PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland